CLINICAL TRIAL: NCT05985603
Title: Comparison of Mirror Therapy and Modified Constrain Induced Movement Therapy on Risk of Fall, Balance and Gait in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01665 Bakhtawar Tariq
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Stroke
Keywords: CIMT; Mirror Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIMT Group (Experimental): In this group of patients CIMT technique will be used for treatment
  Interventions: Other: CIMT Group
- Mirror Therapy Group (Experimental): patient will perform movements in semi-reclined and sitting positions with the mirror placed between the two lower extremities.
  Interventions: Other: Mirror Therapy group

INTERVENTIONS:
Other: CIMT Group — In this group of patients CIMT technique will be used for treatment
  Arms: CIMT Group
Other: Mirror Therapy group — patient will perform movements in semi-reclined and sitting positions with the mirror placed between the two lower extremities.
  Arms: Mirror Therapy Group

SUMMARY:
There will be a difference between modified constraint induced movement therapy and Mirror Therapy on lower limb for risk of fall, balance and gait in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* A Hemiplegia due to unilateral stroke
* Sub-acute and chronic stroke
* Stroke survivors between 21 and 70 years old will be recruited
* Both genders
* NIH Stroke scale below 20
* Mini-Mental State Examination above 24
* Function in Sitting Test (FIST) above 42/56

Exclusion Criteria:

* Patients with depression who will be unable to cooperate during treatment
* Patients who cannot perform the active movement of limb due to prestroke muscoskeletal problems
* Cardiopulmonary diseases which could hinder their ability to participate in rehabilitation
* Spasticity of Modified Ashworth Scale (MAS) II or higher
* Patients with Any neuron disease and Patients with lower-limb impairment caused by other neurological diseases or inability to comply with study protocol will be excluded.
* Visual and auditory abnormalities

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
NIH Stroke Scale - NIHSS | 2,4,8 week
  It comprises of 15 items with each having responses scored on a 0-4 points scale. The overall score ranges from 0-42 points with higher scores specifying pronounced neurological deficits
Mini-mental state examination | 2,4,8 week
  Cognitive status by the mini-mental state examination (mmse)Mini-Mental State Examination (MMSE) is a tool that can quickly diagnose if a person suffers from mild cognitive impairment (MCI) through answering questions in different cognitive domains. The MMSE demonstrates moderately high levels of reliability. It has been reported to be internally consistent
POMA | 2,4,8 week
  After interventions POMA for assessing risk of fall will be used. The POMA is used to examine balance and mobility in the elderly (Tinetti 1986). This examination tool consists of the balance subscale (9 items, 16 points) and gait subscale (8 items, 12 points), totaling 28 points.
Berg balance scale | 2,4,8 week
  A five-point scale, ranging from 0-4. "0" indicates the lowest level of function and "4" the highest level of function. Total Score = 0-56. Score of 41-56 = low fall risk, 21-40 = medium fall risk, 0-20 = high fall risk.
10 Meter walk test / 10mwt | 2,4,8 week
  Calculating Gait Speed - total distance/time. For example: if you did a 10-meter gait speed test and it took you 7 seconds, the equation would like: 10 meters / 7 seconds = 1.4 meters per second. The 10MWT intra-rater and inter-rater reliability were good (ICC between 0.76 until 0.9) and excellent (ICC > 0.9), respectively. The minimal detectable change for intra-rater reliability was 0.188 m/s.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Bashir, MS, Principal Investigator — Riphah International University
Locations (1):
- Helping Hand Institute Of rehabilitation sciences, Mansehra, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oh K, Im N, Lee Y, Lim N, Cho T, Ryu S, Yoon S. Effect of Antigravity Treadmill Gait Training on Gait Function and Fall Risk in Stroke Patients. Ann Rehabil Med. 2022 Jun;46(3):114-121. doi: 10.5535/arm.22034. Epub 2022 Jun 30. PMID 35793900
- [Background] Okonkwo UP, Agbo CF, Ibeneme SC, Igwe ES, Akosile CO, Onwuakagba IU, Emmanuel OC, Maduagwu SM, Ezenwankwo EF, Ekechukwu EN. The Burden and Quality of life of Caregivers of Stroke Survivors with Cognitive Impairment in Selected Healthcare Facilities in Anambra State, Nigeria. Gerontol Geriatr Med. 2022 Sep 27;8:23337214221126329. doi: 10.1177/23337214221126329. eCollection 2022 Jan-Dec. PMID 36189374
- [Background] Wagatsuma M, Kim T, Sitagata P, Lee E, Vrongistinos K, Jung T. The biomechanical investigation of the relationship between balance and muscular strength in people with chronic stroke: a pilot cross-sectional study. Top Stroke Rehabil. 2019 Apr;26(3):173-179. doi: 10.1080/10749357.2019.1574417. Epub 2019 Feb 11. PMID 30741610
- [Background] Khan F, Abusharha S, Alfuraidy A, Nimatallah K, Almalki R, Basaffar R, Mirdad M, Chevidikunnan MF, Basuodan R. Prediction of Factors Affecting Mobility in Patients with Stroke and Finding the Mediation Effect of Balance on Mobility: A Cross-Sectional Study. Int J Environ Res Public Health. 2022 Dec 10;19(24):16612. doi: 10.3390/ijerph192416612. PMID 36554493
- [Background] Li J, Zhong D, Ye J, He M, Liu X, Zheng H, Jin R, Zhang SL. Rehabilitation for balance impairment in patients after stroke: a protocol of a systematic review and network meta-analysis. BMJ Open. 2019 Jul 19;9(7):e026844. doi: 10.1136/bmjopen-2018-026844. PMID 31326927
- [Background] Arienti C, Lazzarini SG, Pollock A, Negrini S. Rehabilitation interventions for improving balance following stroke: An overview of systematic reviews. PLoS One. 2019 Jul 19;14(7):e0219781. doi: 10.1371/journal.pone.0219781. eCollection 2019. PMID 31323068
- [Background] Herrador Colmenero L, Perez Marmol JM, Marti-Garcia C, Querol Zaldivar MLA, Tapia Haro RM, Castro Sanchez AM, Aguilar-Ferrandiz ME. Effectiveness of mirror therapy, motor imagery, and virtual feedback on phantom limb pain following amputation: A systematic review. Prosthet Orthot Int. 2018 Jun;42(3):288-298. doi: 10.1177/0309364617740230. Epub 2017 Nov 20. PMID 29153043
- [Background] Ju Y, Yoon IJ. The effects of modified constraint-induced movement therapy and mirror therapy on upper extremity function and its influence on activities of daily living. J Phys Ther Sci. 2018 Jan;30(1):77-81. doi: 10.1589/jpts.30.77. Epub 2018 Jan 27. PMID 29410571
- [Background] Garrido M M, Alvarez E E, Acevedo P F, Moyano V A, Castillo N N, Cavada Ch G. Early transcranial direct current stimulation with modified constraint-induced movement therapy for motor and functional upper limb recovery in hospitalized patients with stroke: A randomized, multicentre, double-blind, clinical trial. Brain Stimul. 2023 Jan-Feb;16(1):40-47. doi: 10.1016/j.brs.2022.12.008. Epub 2022 Dec 28. PMID 36584748
- [Background] E Silva EMGS, Ribeiro TS, da Silva TCC, Costa MFP, Cavalcanti FADC, Lindquist ARR. Effects of constraint-induced movement therapy for lower limbs on measurements of functional mobility and postural balance in subjects with stroke: a randomized controlled trial. Top Stroke Rehabil. 2017 Dec;24(8):555-561. doi: 10.1080/10749357.2017.1366011. Epub 2017 Aug 31. PMID 28859603
- [Background] Wang D, Xiang J, He Y, Yuan M, Dong L, Ye Z, Mao W. The Mechanism and Clinical Application of Constraint-Induced Movement Therapy in Stroke Rehabilitation. Front Behav Neurosci. 2022 Jun 21;16:828599. doi: 10.3389/fnbeh.2022.828599. eCollection 2022. PMID 35801093
- [Background] Yoon JA, Koo BI, Shin MJ, Shin YB, Ko HY, Shin YI. Effect of constraint-induced movement therapy and mirror therapy for patients with subacute stroke. Ann Rehabil Med. 2014 Aug;38(4):458-66. doi: 10.5535/arm.2014.38.4.458. Epub 2014 Aug 28. PMID 25229024
- [Background] Kim K, Lee S, Kim D, Lee K, Kim Y. Effects of mirror therapy combined with motor tasks on upper extremity function and activities daily living of stroke patients. J Phys Ther Sci. 2016 Jan;28(2):483-7. doi: 10.1589/jpts.28.483. Epub 2016 Feb 29. PMID 27065534